CLINICAL TRIAL: NCT02612064
Title: A Clinical Study Investigating the Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Brief Title: The Efficacy of an Occluding Dentifrice in Providing Relief From Dentinal Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 205072
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stannous Fluoride dentifice (Experimental): Participants will apply (under supervision) a pea-sized dose of experimental dentifrice containing 0.454% w/w stannous fluoride (1100ppm) to each of the two qualifying teeth using their finger by direct application and gently rubbing into the tooth's cervical margin for the allocated time. No rinsing will be permitted
  Interventions: Device: Stannous Fluoride dentifice
- Sodium Monofluorophosphate dentifrice (Other): Participants will apply (under supervision) a pea-sized dose of dentifrice containing Dentifrice containing 0.76% sodium monofluorophosphate (1000ppm fluoride)to each of the two qualifying teeth using their finger by direct application and gently rubbing into the tooth's cervical margin for the allocated time. No rinsing will be permitted.
  Interventions: Other: Sodium Monofluorophosphate dentifrice

INTERVENTIONS:
Device: Stannous Fluoride dentifice — Experimental dentifrice containing 0.454% w/w stannous fluoride (1100ppm)
  Arms: Stannous Fluoride dentifice
Other: Sodium Monofluorophosphate dentifrice — Dentifrice containing 0.76% sodium monofluorophosphate (1000ppm fluoride)
  Arms: Sodium Monofluorophosphate dentifrice

SUMMARY:
This single centre, dual site, comparative design study will be used to investigate the efficacy of an experimental stannous fluoride containing dentifrice in relieving dentinal hypersensitivity (DH) after short term use

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee:

A. No clinically significant and relevant abnormalities in medical history or upon oral examination.

B. Absence of any condition that would impact on the participant's safety or wellbeing or affect the individual's ability to understand and follow study procedures and requirements.

- Dental health

At Screening:

A. Self-reported history of dentinal hypersensitivity (DH) lasting more than six months but not more than 10 years.

B. Good general oral health, with a minimum of 20 natural teeth.

C. Minimum of 2 accessible non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, that meet all of the following criteria:

* Signs of facial/cervical gingival recession and/or signs of erosion or abrasion (EAR).
* Tooth with modified gingival index (MGI) score =0 adjacent to the test area (exposed dentine) only and a clinical mobility of ≤1.
* Tooth with signs of sensitivity measured by qualifying evaporative air assessment (Y/N response).

At Baseline:

D. Minimum of two, non-adjacent accessible teeth (incisors, canines, pre-molars), that meet all of the following criteria:

- Tooth with signs of sensitivity, measured by qualifying tactile stimulus (Yeaple ≤ 20g) and evaporative air assessment (Schiff Sensitivity Score ≥ 2)

Exclusion Criteria:

* Pregnant or breast feeding women
* Daily doses of medication/treatments which, in the opinion of the investigator, could interfere with the perception of pain.
* Currently taking antibiotics or has taken antibiotics within two weeks of Baseline.
* Daily dose of a medication which, in the opinion of the investigator, is causing xerostomia. - Presence of chronic debilitating disease which, in the opinion of the investigator, could affect study outcomes.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit.
* Recent history (within the last year) of alcohol or other substance abuse
* Dental prophylaxis within four weeks of Screening.
* Tongue or lip piercing or presence of dental implants.
* Desensitizing treatment within eight weeks of Screening (professional sensitivity treatments and non-toothpaste sensitivity treatments).
* Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of Screening, scaling or root planning within 3 months of Screening.
* Teeth bleaching within eight weeks of Screening
* Tooth with evidence of current or recent caries, or reported treatment of decay within 12 months of Screening.
* Tooth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns or veneers, orthodontic bands or cracked enamel. Sensitive teeth with contributing aetiologies other than erosion, abrasion or recession of exposed dentine.
* Sensitive tooth not expected to respond to treatment with an over-the-counter toothpaste in the opinion of the investigator.
* Use of an oral care product indicated for the relief of dentine hypersensitivity within eight weeks of screening
* Individuals who require antibiotic prophylaxis for dental procedures

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 488 (Actual)
Dates: Start 2015-11-01; Primary Completion 2016-06-03 (Actual); Study Completion 2016-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Ellesmere Port, Cheshire
  - GSK Investigational Site, Metropolitan Borough of Wirral

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site in United Kingdom (UK).
Pre-assignment Details: In total, 488 participants were screened, out of which 230 participants were randomized.
Groups:
- Stannous Fluoride: Test: Participants were instructed to apply a pea-sized dose of experimental dentifrice containing 0.454% w/w stannous fluoride (1100 ppm fluoride) to each of the two qualifying teeth using their finger by direct application and gently rubbing into the tooth's cervical margin for the allocated time. No rinsing was permitted after direct application with treatment. For at home use, participants then brushed their whole mouth for at least 1 minute and were permitted to rinse with 5ml tap water (room temperature) for 5 seconds maximum after brushing.
- Sodium Monofluorophosphate: Control: Participants were instructed to apply a pea-sized dose of dentifrice containing 0.76% w/w sodium monofluorophosphate (1000 ppm fluoride) to each of the two qualifying teeth using their finger by direct application and gently rubbing into the tooth's cervical margin for the allocated time. No rinsing was permitted after direct application with treatment. For at home use, participants then brushed their whole mouth for at least 1 minute and were permitted to rinse with tap water.
Period: Overall Study
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Started | 115 | 115
Completed | 114 | 112
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate | Total
Number analyzed (Participants) | 115 | 115 | 230
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.7 (8.62) | 39.9 (9.18) | 40.3 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 24 | 23 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 115 | 115 | 230
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 112 | 112 | 224
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Schiff Sensitivity Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — Assessed by examiner as participant's response to an evaporative (air) stimulus after stimulation of each individual tooth, scored using Schiff sensitivity scale range of 0-3; 0=Participant does not respond to air stimulation; 1=Participant responds to air stimulus but does not request discontinuation of stimulus; 2=Participant responds to air stimulus & requests discontinuation or moves from stimulus; 3=Participant responds to stimulus, considers stimulus to be painful, & requests discontinuation of stimulus. A reduction in Schiff Sensitivity score indicates improvement in sensitivity. Population: Analysis for this outcome was performed on intent-to-treat (ITT) population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
  score on a scale | 2.82 (0.333) | 2.80 (0.330) | 2.81 (0.331)
Tactile Sensitivity - Tactile Threshold at Baseline [Mean (Standard Deviation); unit: gram (g)] — Tactile threshold was assessed by examiner using a constant pressure probe (Yeaple probe) which allowed application of a known force to the dentin surface from 10 g to an upper threshold of 80g in increments of 10g. Tactile threshold is the maximum pressure applied at which participant do not report any pain or discomfort. Tactile threshold for each tooth was determined by asking participant whether sensation caused discomfort. The pressure setting at which participant gave two consecutive 'yes' responses was recorded as tactile threshold. Higher tactile threshold, less sensitive tooth. Population: Analysis for this outcome was performed on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
  gram (g) | 12.26 (2.905) | 12.52 (3.202) | 12.39 (3.053)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Schiff Sensitivity Score on Day 3
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows - 0: Participant does not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score was indicative of an improvement in sensitivity.
Time Frame: Baseline to 3 days
Population: Analysis for this outcome was performed on ITT population, defined as all participants who were randomized, received the study treatment at least once and provided at least one post-baseline (post treatment) assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 115 | 115
Score on a scale | -0.96 (1.003) | -0.77 (0.947)
Statistical Analysis 1: Comparison: Stannous Fluoride vs Sodium Monofluorophosphate; All statistical analyses were conducted under the null hypothesis (H0) of no difference between treatments versus the alternate hypothesis (H1) of a difference between treatments; Test type: Superiority or Other; p = 0.1575, ANCOVA; Change from baseline in Schiff Sensitivity Score as response, treatment as a factor and baseline Schiff sensitivity as a covariate; Least Square (LS) mean difference = -0.18, 95% CI 2-sided [-0.442 to 0.072] — Difference is first named dentifrice minus second named dentifrice such that a negative difference favours first named dentifrice

2. Secondary Outcome: Change From Baseline in Schiff Sensitivity Score Post First Treatment by Direct Application
Description: The examiner assessed the participant's response to an evaporative air stimulus for each tooth using the Schiff Sensitivity Scale which was scored as follows 0: Participant does not respond to air stimulation; 1: Participant responded to air stimulus but does not request discontinuation of stimulus; 2: Participant responded to air stimulus and requests discontinuation or moves from stimulus; 3: Participant responded to stimulus, considered stimulus to be painful, and requested discontinuation of the stimulus. A reduction in Schiff Sensitivity score was indicative of an improvement in sensitivity.
Time Frame: Baseline to 60 seconds post first treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 115 | 115
score on a scale | -0.41 (0.760) | -0.31 (0.690)

3. Secondary Outcome: Change From Baseline in Tactile Threshold Post First Treatment by Direct Application and on Day 3
Description: The examiner assessed the response to tactile sensitivity using a Yeaple probe which allowed application of a known force to the dentin surface, starting at 10g and rising in increments of 10g until the tactile threshold or maximum force was reached. The tactile threshold for each tooth was determined by asking the participant whether the sensation caused discomfort. The pressure setting at which the participant gives two consecutive 'yes' responses was recorded as the tactile threshold. The higher the tactile threshold, the less sensitive the tooth. At baseline, the maximum force used was 20g; at all subsequent visits, it was 80g.
Time Frame: Baseline, 60 seconds post first treatment, Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
Number analyzed (Participants) | 115 | 115
g
  Change from Baseline to Day 0, Post-Treatment | 8.83 (16.254) | 4.74 (9.975)
  Change from Baseline to Day 3 | 15.09 (20.642) | 12.77 (19.543)

ADVERSE EVENTS:
Arm/Group | Stannous Fluoride | Sodium Monofluorophosphate
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/115
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/115
Other Adverse Events (participants affected / at risk) | 3/115 | 5/115
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stannous Fluoride (N=115) | Sodium Monofluorophosphate (N=115)
Chapped Lips (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.